CLINICAL TRIAL: NCT05063955
Title: Socioeconomic Factors and Mechanisms of Sarcopenia and Muscle Strength in Chronic Heart Failure Patients
Brief Title: Mechanism of Sarcopenia in Heart Failure
Acronym: MUSCLE-CHF
Status: Recruiting | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Henrik Wiggers, Professor, Aarhus University Hospital
Other Study IDs: 73789
Record Dates: First submitted 2021-06-01; First posted 2021-10-01 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Heart Failure; Sarcopenia; Cachexia
Keywords: Heart failure; Sarcopenia; Cachexia
MeSH Terms: conditions — Heart Failure; Sarcopenia; Cachexia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Heart Failure: Patients with heart failure with preserved, mid-range or reduced ejection fraction (NYHA I-IV) according to European Society of Cardiology guidelines.
- Controls: Age and sex matched control group. Individuals with no history of cardiovascular disease or severe lung, musculoskeletal or neurological disease.

SUMMARY:
The aim of the study is to provide information on the interaction between socioeconomic factors, daily physical activity, nutrition and lifestyle on loss of muscle mass and muscle function in patients with heart failure.

DETAILED DESCRIPTION:
A total of 200 consecutive heart failure patients will be included and 50 age and sex-matched individuals with no history of cardiovascular disease will serve as controls.

Baseline variables of body composition, physical capacity, daily physical activity, nutritional status, quality of life, socioeconomic status and insulin resistance will be obtained along with a skeletal muscle tissue biopsy and blood samples for laboratory analyses.

Baseline variables from heart failure patients will be compared to healthy controls.

Patients and controls will be invited to follow-up visits at 12 and 36 months. Changes in baseline variables will be analyzed.

Events will be identified through national registries.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide valid informed consent.
2. Heart failure with preserved, mid-range or reduced ejection fraction (NYHA I-IV) according to European Society of Cardiology guidelines.

Exclusion Criteria:

1. Cancer requiring treatment (e.g. prostate cancer on watchful waiting does not exclude patients).
2. Severe musculoskeletal or neurological disability.
3. Severe lung disease with a forced expiratory volume 1 < 40% of predicted. Treatment with anticoagulants (warfarin, apixaban, edoxaban, dabigatran and rivaroxaban) is an exclusion criterion for muscle biopsy. Patients with anticoagulant treatment will be invited to participate in the study without muscle biopsy.
4. Other comorbidities that prevent the patient from participating in the study examinations as judged by the investigator.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 200 consecutive heart failure patients will be included and 50 age and sex matched individuals with no history of cardiovascular disease will serve as controls.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-12-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical performance, peak VO2 | From baseline to 12 and 36 months
  Change in peak oxygen uptake (peak VO2), measured in ml O2/kg/min
Physical performance, walking distance | From baseline to 12 and 36 months
  Change in walking distance (6MWT) in meters
Physical performance, muscle strength | From baseline to 12 and 36 months
  Change in knee extension/flexion isokinetic strength (assessed by peak torque, Nm) and isometric strength (assessed by peak torque, Nm)

SECONDARY OUTCOMES:
Cardiovascular events | During follow-up of 10 years
  Incidence of a composite endpoint of death, hospitalization with worsening of heart failure other cardiovascular events (myocardial infarction, unstable angina, revascularization and stroke) and non-cardiovascular hospitalizations
Body composition | From baseline to 12 and 36 months
  Change in appendicular lean mass (measured in grams) and fat mass (measured in grams)
Muscle tissue fiber types | From baseline to 12 and 36 months
  Change in ratio between muscle fiber types (type I, IIa and IIb) assessed by immunohistochemistry
Muscle tissue cellular composition | From baseline to 12 and 36 months
  Change in muscle tissue cellular composition assessed by cell sorting
Muscle tissue mitochondrial function | From baseline to 12 and 36 months
  Change in muscle mitochondrial function assessed by high-resolution respirometry
Daily physical activity | From baseline to 12 and 36 months
  Change in daily physical activity assessed by 7-day accelerometry
Insulin resistance | From baseline to 12 and 36 months
  Changes in insulin resistance assessed by Homeostatic Model Assessment for Insulin Resistance (HOMA-IR)
Whole body metabolism | From baseline to 12 and 36 months
  Changes in circulating metabolic markers
Muscle metabolism | From baseline to 12 and 36 months
  Changes in metabolic signature of muscle tissue assessed by liquid chromatography-high-resolution mass spectrometry
Symptoms | From baseline to 12 and 36 months
  Changes in the Minnesota Living with Heart Failure Questionnaire score (range 0-105, from best to worst)

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Wiggers, Prof., Study Chair — Aarhus University Hospital; Andreas B Tinggaard, MD, Study Chair — Aarhus University Hospital; Søren P Johnsen, Prof., Study Chair — Aalborg University Hospital; Helene Nørrelund, Ass. Prof., Study Chair — Aarhus University Hospital; Anders H Larsen, MD, PhD, Study Chair — Aarhus University Hospital; Peter Leutscher, Prof., Study Chair — Regionshospital Nordjylland; Peter B Stæhr, MD, PhD, Study Chair — Regionshospital Nordjylland; Steen H Jørgensen, MD, Study Chair — Regionshospital Nordjylland; Niels Jessen, Prof., Study Chair — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tinggaard AB, Sorensen L, Vissing K, Jessen N, Norrelund H, Wiggers H. Daily physical activity and prognostic implications in patients with heart failure: an accelerometer study. Clin Res Cardiol. 2025 May;114(5):616-628. doi: 10.1007/s00392-024-02508-0. Epub 2024 Sep 2. PMID 39222281